# Effects of FDA Authorized Smokeless Tobacco Claims among US Adults who Smoke Cigarettes

NCT Number: NCT06927700

Informed Consent Document

Document Date: April 3, 2025

Protocol Title: Effects of FDA Authorized Smokeless Tobacco Claims

Version Date: v3, 4/3/25

#### **CONSENT TO TAKE PART IN A RESEARCH STUDY**

**TITLE OF STUDY**: Perceptions of tobacco product ads and messages

Principal Investigator: Olivia Wackowski, PhD, MPH

This online consent form is part of an informed consent process for a research study and it will provide information that will help you decide whether you want to take part in the study. It is your choice to take part or not. Ask questions if there is anything in the form that is not clear to you. If you decide to take part, instructions at the end of page will tell you what to do next. Your alternative to taking part in the research is not to take part in it.

### Who is conducting this research study and what is it about?

You are being asked to take part in research conducted by Olivia Wackowski, PhD, who is an Associate Professor in the Institute for Nicotine & Tobacco Studies at Rutgers University. The study will help researchers understand people's interest in different tobacco products and reactions to advertisements and information about these products.

### What will I be asked to do if I take part?

You will answer questions about your experience with tobacco products and your opinions of tobacco ads and products you will see in the survey. The survey will take about 10 minutes to complete.

### What are the risks and/or discomforts I might experience if I take part in the study?

We will not ask sensitive questions and no risks are expected. As with all Ipsos KnowledgePanel® surveys, responding to this survey, or to any individual question on the survey, is completely voluntary. Your responses remain anonymous to us and will be used for research analyses only.

## Are there any benefits to me if I choose to take part in this study?

There are no direct benefits to you for taking part in this research. Your answers will help regulators, researchers and professionals in decision making about different types of tobacco ads and messages.

#### Will I be paid to take part in this study?

You will be compensated based on your agreement with Ipsos.

## How will information about me be kept private or confidential?

All efforts will be made to keep your responses confidential, but total confidentiality cannot be guaranteed. Ipsos will collect and forward your deidentified responses to us. We will not receive any information that can identify you. We will download your responses to a secure file that requires a password to access. Only study staff will have access to the password. No information that can identify you will appear in any professional presentation or publication.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH). This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that

Protocol Title: Effects of FDA Authorized Smokeless Tobacco Claims

Version Date: v3, 4/3/25

federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

## What will happen to information I provide in the research after the study is over?

A final dataset with all participants' responses to this survey will be made publicly available on a data repository website. As such, responses may be used or distributed to investigators for other research without obtaining additional informed consent from you. However, it will not include any information that can identify you. Your participation is anonymous.

## What will happen if I do not want to take part or decide later not to stay in the study?

Your participation is voluntary. If you choose to take part now, you may change your mind and withdraw once you start the survey. In addition, you can choose to skip questions that you do not wish to answer. If you do not click on the 'submit' button after completing the form, your responses will not be recorded. However, once you click the 'submit' button at the end of the form, your responses cannot be withdrawn as we will not know which ones are yours.

### Who can I call if I have questions?

If you have questions about taking part in this study, you can contact the Principal Investigator: Olivia Wackowski, <u>olivia.wackowski@rutgers.edu</u>. If you have questions about your rights as a research subject, you can contact the IRB Director at: (732) 235-9806 or the Rutgers Human Research Protection Program at (973) 972-1149 or email <u>IRBOffice@research.rutgers.edu</u>. You may also contact the Ipsos KnowledgePanel Member Support at 1-800-782-6899.

Please print out this consent form if you would like a copy of it for your files.

By beginning this research, I acknowledge that I am 21 years of age or older and have read and understand the information. I agree to take part in the research, with the knowledge that I am free to withdraw my participation in the research without penalty.

If you consent to participate in this study, please click the NEXT button below to begin the survey.

Protocol Title: Effects of FDA Authorized Smokeless Tobacco Claims

Version Date: v3, 4/3/25